CLINICAL TRIAL: NCT00208598
Title: Measures of Obesity and Co-Morbid Conditions in Maori
Status: Completed | Type: Observational
Sponsor: Edgar National Centre for Diabetes Research (Other)
Other Study IDs: ENCDR_3
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Body Composition
Keywords: Maori; Body Composition; DEXA; Cardiovascular disease; Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
It has been proposed that a higher cut off for BMI (body mass index) is to be used in Maori to define overweight and obesity. However, no one has assessed the prevalence of co-morbid conditions associated with BMI. It is well known that Maori are at greater risk of diabetes and cardiovascular disease compared to non-Maori and a delay in the identification of those who are overweight and obese may be detrimental for Maori. We will assess BMI, other measures of adiposity and prevalence of co-morbid conditions with a comparison with a similar matched non-Maori population.

DETAILED DESCRIPTION:
This is a body composition analysis study of people self-identifying Maori and non-Maori participants from both Dunedin and Invercargill. The study consists of a clinical visit for anthropometry and oral glucose tolerance test (OGTT), followed by a single Dexa Scan visit. Participants meeting all the inclusion criteria were invited to participate in the study.

Outcome will be determined by examining Dexa Scan data and surrogate clinical endpoints. The clinical endpoints include: anthropometric measurements, Dexa analysis, bioelectric impedance, and BP measurements, and the biochemical measures of: lipid profile, fasting insulin and glucose, liver functions and uric acid levels.

ELIGIBILITY:
Inclusion Criteria:

* Self identify as Maori and non-Maori aged between 18-68 years
* Male and female
* Non-diabetic
* Resident of Dunedin and Invercargill

Exclusion Criteria:

* The presence of diabetes, renal or liver failure, or any other medical condition which is unstable and for which they are currently having active treatment

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2003-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Jim I Mann, FRACP, PhD, Study Director — Edgar National Centre for Diabetes Research
Locations (1):
- Edgar National Centre for Diabetes Research, Dunedin, Otago, New Zealand

REFERENCES:
- See also: Edgar National Centre for Diabetes Research, NZ website — http://www.otago.ac.nz/diabetes